CLINICAL TRIAL: NCT05064657
Title: The Effect of Two Different Applications on Reducing Pain and Fear During Draw Blood From Children
Brief Title: The Effect of Two Method to Reducing Pain and Fear During Draw Blood From Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Fatma Taş Arslan, Professor, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SelcukU-01-2020
Record Dates: First submitted 2021-06-29; First posted 2021-10-01 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Pain, Procedural; Pain Management; Child, Only
Keywords: pain; procedural; fear; child; distraction methods
MeSH Terms: conditions — Pain, Procedural; Agnosia; Pain

STUDY DESIGN:
Intervention Model Description: Parallel Assignment First sub purpose was designed as parallel group, two intervention groups in pre-test and post-test order, and a randomized controlled control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Group (Experimental): Experimental Group (ball squeezing) The group were used a ball squeezing method during the blood collection process.
  The children were given a ball during the blood draw and told to tighten and loosen it.
  Interventions: Procedure: Bubble blowing method
- Active Comparator (Active Comparator): Active Comparator ( bubble blowing) The group were used a bubble blowing method during the blood collection process. During the blood collection process, the children were asked to blow bubbles by giving the apparatus inside the foam bubble to their free arm.
  Interventions: Procedure: Bubble blowing method
- Control Group (No Intervention): No intervention

INTERVENTIONS:
Procedure: Bubble blowing method — The investigators were used "Bubble blowing method" and "ball squeezing method".
  To child were used a ball squeezing method during the blood collection process.
  Other Names: Ball squeezing method
  Arms: Active Comparator; Experimental Group

SUMMARY:
This study was conducted to evaluate the effects of two different distraction methods on reducing pain and fear during blood collection from children.

The study was conducted between January 2020 and May 2021.

DETAILED DESCRIPTION:
The study was a pretest-posttest, parallel group randomized controlled experimental design.

H0: The pain and fear mean scores of the intervention group, in which the distraction method (ball squeezing and blowing bubbles) was applied during the blood collection process, was not different from the control group.

The study was carried out with the participation of 111 children aged 6-12 years and their parents, who underwent blood collection in the emergency department of a state hospital.

Children were randomly assigned to blowing bubbles (n:37), ball squeezing (n:37) and control (n:37) groups. Bubble blowing and ball squeezing methods were used to distract attention during the blood collection process. Data were collected with Child and Family Information Form, Wong Baker Faces Pain Scale, Child Fear Scale. Pretest and posttest measurements were recorded separately by the child, parent and researcher. Descriptive statistics, Chi-square test, one-way analysis of variance, Tamhane's T2 test, t test for dependent groups were used in the analysis of the data. The statistical significance of the results was taken as p<0,05

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 6-12
* The child's willingness to voluntarily participate in the study
* Parent's willingness to participate in the study voluntarily
* Parent and child can speak Turkish

Exclusion Criteria:

* The child has a disease that causes chronic pain
* The child has a hearing or visual impairment
* The child has a mental or neurological disability
* The child has used drugs that will create an analgesic effect in the last 24 hours before the application

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 111 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Wong Baker Pain Faces Scale mean score | First ten minute
  Wong-Baker Pain Faces Scale is widely used with people ages three and older, not limited to children. This self-assessment tool must be understood by the patient, so they are able to choose the face that best illustrates the physical pain they are experiencing. It is a tool to be used by a third person, parents, healthcare professionals, or caregivers, to assess the patient's pain. The scale is 0-10 scale. The six illustrated faces on the cards show a range of emotions, from a smiling face (0 'no pain) to a crying face (10 "worst pain"). 0 indicates no pain, 10 indicates the most severe pain. It defines the child's pain level before and after the blood collection.
Children's Fear Scale mean score | First ten minute
  Children's Fear Scale is a scale of 0-4 showing five faces ranging from a neutral expression (0 = no concern) to the feared face (4 = severe anxiety). A score of 0 indicates no fear and a score of 4 indicates extremely fearful. Defines the change of fear level before and after during the blood collection.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Tas Arslan, Prof., Study Director — Selcuk University; Neşe Oluç, Msc, Principal Investigator — Selcuk University
Locations (1):
- Selcuk University, Konya, Selcuklu, Turkey (Türkiye)

REFERENCES:
- [Derived] Oluc N, Tas Arslan F. The effect of two different methods on reducing the pain and fear during phlebotomy to children: A randomized controlled trial. Int Emerg Nurs. 2024 Feb;72:101386. doi: 10.1016/j.ienj.2023.101386. Epub 2023 Nov 18. PMID 37984025